CLINICAL TRIAL: NCT00413959
Title: Phase II Study Investigating the Efficacy of VELCADE®, Rituximab, Cyclophosphamide and Decadron (VRCD Regimen) in Front-line Therapy of Patients With Low-grade Non-Hodgkin's Lymphoma
Brief Title: VELCADE,Rituximab,Cyclophosphamide and Decadron
Acronym: VRCD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Oncology Specialists, S.C. (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Director of Research, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0606
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, B-Cell
Keywords: NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Bortezomib; Rituximab; Cyclophosphamide; Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velcade, Rituximab,Cyclophosphamide & Decadron (Experimental): Velcade 375 mg/m^2 given intravenously on days 1, 8, 15 and 22 during the first cycle then on day 1 of each subsequent cycle.
  Interventions: Drug: VELCADE®; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Decadron

INTERVENTIONS:
Drug: VELCADE® — 1.6 mg/m^2 of Velcade® given intravenously on days 1, 8, 15 and 22.
  Other Names: Bortezomib
Drug: Rituximab — 375 mg/m^2 of Rituximab given intravenously on days 1, 8, 15 and 22 during the first cycle then on day 1 of each subsequent cycle.
  Other Names: Rituxan
Drug: Cyclophosphamide — 400 mg/m^2 of Cyclophosphamide given orally on days 1-4 of each cycle.
  Other Names: Cytoxan
Drug: Decadron — 40 mg given orally on days 1, 2, 8, 9, 15, 16, 22 and 23
  Other Names: dexamethasone

SUMMARY:
Overall response rate and Time to disease progression using this regimen in patients with low-grade B-Cell Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
This is a phase II open label study that is looking at the VRCD combination regimen in patients with previously untreated low-grade Non-Hodgkin's Lymphoma. Treatment will start by combining oral dexamethasone and cyclophosphamide with intravenous VELCADE, rituximab. Chemotherapy cycles will be given as outlined below every 35-days and will continue until two cycles beyond complete remission (CR), toxicity, patient's withdrawal, disease progression, or a maximum of 8 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Small Lymphocytic Lymphoma
* Follicular Cell Lymphoma (grades I and II)
* Mantle Cell Lymphoma patients that are not considered eligible for high-dose therapy and stem cell transplant
* Lymphoplasmacytic lymphoma including Waldenstrom's Macroglobulinemia
* Marginal Zone Lymphoma
* MALT Lymphoma that has ONLY failed antibiotic therapy or involved field radiation.
* Adequate bone marrow function, renal function, and hepatic function as outlined in details below.
* ECOG performance status of 0, 1, or 2
* Able to read, understand, and sign an IRB approved informed consent

Exclusion Criteria:

* Known HIV positive status
* Known CNS involvement
* Prior therapy for lymphoma EXCLUDING antibiotic treatment for MALT-Type NHL.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, SC
Locations (2):
- United States (2):
  - Onocology Specialists, S.C, Niles, Illinois
  - Oncology Specialists, S.C, Park Ridge, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Rituximab (R) are alone or R based chemo programs are front line approach LG-NHL pts requiring therapy. Identifying programs that are effective in the elderly pts is challenging. These pts were recruited in our private practice.
Pre-assignment Details: Eligible pts had LG-NHL requiring treatment. Mantel cell NHL pts who were'nt transplant eligible and MALToma pts who failed RT and antibiotics were allowed.
Period: Overall Study
Arm/Group | Velcade, Rituximab,Cyclophosphamide & Decadron
Started | 12
Completed | 11
Not Completed | 1
Not completed — Pt had only one cycle. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Velcade, Rituximab,Cyclophosphamide & Decadron
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Using This Regimen in Patients With Low-grade B-Cell Non-Hodgkin's Lymphoma.
Description: Percentage of complete responders plus percentage of partial responders equals overall response rate.
Time Frame: 4 years
Population: 1 pt withdrew before completing two cycles and was not evaluable for OS.
Measure: Number; unit: percentage of patients
Arm/Group | Velcade, Rituximab,Cyclophosphamide & Decadron
Number analyzed (Participants) | 11
percentage of patients | 90

2. Secondary Outcome: Overall Survival
Description: The study was closed prematurely due to slow accrual. When the study closed only two patients had died, making the OS 83%.
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Velcade, Rituximab,Cyclophosphamide & Decadron
Number analyzed (Participants) | 11
percentage of participants | 83

ADVERSE EVENTS:
Arm/Group | Velcade, Rituximab,Cyclophosphamide & Decadron
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade, Rituximab,Cyclophosphamide & Decadron (N=12)
Congestive Heart Failure (Cardiac disorders) | 1
Cerebral Vascular Accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade, Rituximab,Cyclophosphamide & Decadron (N=12)
Anxiety Grade 1 & 2 (General disorders) | 2
Abdominal Pain Grade 1 & 2 (Gastrointestinal disorders) | 1
Appetite Decreased Grade 1 & 2 (Gastrointestinal disorders) | 1
Bilirubin Increased Grade 1 & 2 (Renal and urinary disorders) | 1
Alopecia Grade 1 & 2 (General disorders) | 1
Creatinine Increased Grade 1 & 2 (Renal and urinary disorders) | 1
Constipation Grade 1 & 2 (Gastrointestinal disorders) | 1
Cough Grade 1 & 2 (Respiratory, thoracic and mediastinal disorders) | 1
Chills Grade 1 & 2 (General disorders) | 2
Edema Grade 1 & 2 (General disorders) | 2
Fever Grade 1 & 2 (General disorders) | 1
Fatigue Grade 1 & 2 (General disorders) | 4
Hyponatremia Grade 1 & 2 (Gastrointestinal disorders) | 1
Hypertension Grade 1 & 2 (Cardiac disorders) | 1
Hyperglycemia Grade 1 & 2 (Gastrointestinal disorders) | 2
Insomnia Grade 1 & 2 (General disorders) | 1
Leukopenia Grade 1 & 2 (Blood and lymphatic system disorders) | 2
Rash Grade 1 & 2 (Skin and subcutaneous tissue disorders) | 1
Nausea Grade 1 & 2 (Gastrointestinal disorders) | 3
Mucositis Grade 1 & 2 (Gastrointestinal disorders) | 1
Pulmonary Edema Grade 1 & 2 (Respiratory, thoracic and mediastinal disorders) | 1
Nail Changes Grade 1 & 2 (Skin and subcutaneous tissue disorders) | 1
Sweats Grade 1 & 2 (General disorders) | 2
Dry Skin Grade 1 & 2 (Skin and subcutaneous tissue disorders) | 1
Stomatitis Grade 1 & 2 (Gastrointestinal disorders) | 1
Sinus Congestion Grade 1 & 2 (Respiratory, thoracic and mediastinal disorders) | 1
Tronopin Increased Grade 1 & 2 (Blood and lymphatic system disorders) | 1
Triglyceride Increased Grade 1 & 2 (General disorders) | 1
Tongue Swelling Grade 1 & 2 (General disorders) | 1
Weight Decreased Grade 1 & 2 (Gastrointestinal disorders) | 2
Tooth Abcess Grade 1 & 2 (General disorders) | 1
Vomiting Grade 1 & 2 (Gastrointestinal disorders) | 1
Difficulty Walking Grade 1 & 2 (Musculoskeletal and connective tissue disorders) | 2
Chest Pain Grade 3 & 4 (Musculoskeletal and connective tissue disorders) | 1
Hyperglycemia Grade 3 & 4 (Gastrointestinal disorders) | 1
Leukopenia Grade 3 & 4 (Blood and lymphatic system disorders) | 3
Neutropenia Grade 3 & 4 (Blood and lymphatic system disorders) | 3
Orthopnea Grade 3 & 4 (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Edema Grade 3 & 4 (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Emboli Grade 3 & 4 (Respiratory, thoracic and mediastinal disorders) | 1
Shortness of Breath Grade 3 & 4 (Respiratory, thoracic and mediastinal disorders) | 1
Headache Grade 1 & 2 (General disorders) | 1
Pain Grade 1 & 2 (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No